CLINICAL TRIAL: NCT00677599
Title: Reducing Cardiovascular Risk With Dietary Flavonoids in Post Menopausal Women With Type 2 Diabetes
Brief Title: The FLAVO Trial: Dietary Flavonoids and Cardiovascular Disease Risk Reduction in Postmenopausal Women With Type 2 Diabetes
Acronym: FLAVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other); The Bertram Diabetes Centre & Radiology department (Norfolk & Norwich University Hospital, UK) (Unknown); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other); Diabetes UK (Other); Frutarom Netherlands B.V. - Soy producer (Unknown); Barry Callebaut - chocolate manufacturer contracted to produce intervention foods (Unknown)
Responsible Party: Aedin Cassidy; Professor of Nutrition, School of Medicine, Health Policy & Practice, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R15098; REC Ref: 07/H0310/136
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Cardiovascular Disease; Diabetes
Keywords: Cardiovascular disease; type 2 diabetes; flavonoids; cocoa; soy; epicatechin; postmenopausal; carotid intima media thickness; plaque volume
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention A (Active Comparator): Experimental arm enriched with flavonoids
  Interventions: Dietary Supplement: Flavonoid enrichment (cocoa / soy compounds)
- Intervention B (Placebo Comparator)
  Interventions: Dietary Supplement: Flavonoid enrichment (cocoa / soy compounds)

INTERVENTIONS:
Dietary Supplement: Flavonoid enrichment (cocoa / soy compounds) — Flavonoid compounds from cocoa (including epicatechin) and soy to be consumed for 365days in the experimental intervention (versus placebo consumption). 27g chocolate bar the vehicle for flavonoid enrichment.
  Other Names: Flavonoid enrichment of compounds found in cocoa and soy versus placebo control
  Arms: Intervention A
Dietary Supplement: Flavonoid enrichment (cocoa / soy compounds) — 27g placebo chocolate bar to be consumed for 365 days.
  Arms: Intervention B

SUMMARY:
The purpose of this placebo controlled trial is to determine whether a year long intervention with flavonoids (found in cocoa and soy) is more effective in reducing the risk of cardiovascular disease in postmenopausal women with type 2 diabetes, than standard therapy (statins). A range of markers of cardiovascular disease risk are being studied and volunteers are also providing urine and blood samples. 152 postmenopausal women, from the locality, will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria

* Female
* Having had a natural menopause and a minimum of 1 year since last menstruation
* Caucasian
* under 70 years
* Type 2 diabetics
* Those using statins (≥40 mg simvastatin or ≥10 mg atorvastatin) for at least 12 months
* Not currently taking Hormone Replacement Therapy (HRT) and not having taken HRT for a minimum of 6 months prior to commencement
* Having no significant past or present medical history of vascular disease, or cancers (specifically breast, uterine or ovarian)
* Never-smokers, and ex-smokers who have given up smoking at least 12 months before recruitment to the study

Exclusion Criteria

* Currently taking HRT or having taken this medication within 6 months of the trial
* Those prescribed to use statin therapy for less than 12 months Significant past or present medical history of vascular disease (including ECG and enzyme confirmed myocardial infarction, clinical angina, ischaemic stroke peripheral vascular disease, intermittent claudication) or cancer (especially breast, uterine or ovarian)
* Hypertensive's with a systolic BP ≥ 160 mm Hg at maximum, or hypertensive's with a systolic BP ≤160 mm Hg at maximum, but who have received antihypertensive therapy for less than 12 months or have had increases to their medication indicating poor control
* Current smokers or those having given up smoking less than 12 months before recruitment to the study
* Those prescribed aspirin for a period of less than 12 months prior to recruitment
* Those prescribed insulin for a period of less than 12 months prior to recruitment and those having had increases to their medication indicating poor control
* Regular non-prescribed use of anti-inflammatory pain relief medication (i.e. aspirin, paracetamol, cocodamol).
* Taking other counter indicative medication e.g. steroidal medication during the trial, or within 1 month of the trial beginning.
* Taking food / dietary supplements e.g. vitamins, minerals, fish oils, plant oils, isoflavones, soy products, carotenoids during the trial (unless prepared to cease intake during, and 1 month preceding the trial).
* Having vaccinations (excluding the flu vaccination) or antibiotics within 3 months of start of trial, and those with vaccinations scheduled for during the trial
* Parallel participation in another research project which involves dietary intervention and/or sampling of biological fluids/material
* Assessed from the clinical screening: HbA1c ≥ 10%; Creatinine >125µmol/L; ALP > 378 IU/L; ALT >150 IU/L; GGT > 180 IU/L

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular disease risk indictaors - including carotid intima-media thickness (CIMT), total plaque volume (TPV) (at the carotid bifurcation), pulse wave velocity (PWV) and biomarkers of risk in blood samples . | 6 months - 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aedin MM Cassidy, PhD, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia (UK); School of Medicine, Health Policy and Practice, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Curtis PJ, Potter J, Kroon PA, Wilson P, Dhatariya K, Sampson M, Cassidy A. Vascular function and atherosclerosis progression after 1 y of flavonoid intake in statin-treated postmenopausal women with type 2 diabetes: a double-blind randomized controlled trial. Am J Clin Nutr. 2013 May;97(5):936-42. doi: 10.3945/ajcn.112.043745. Epub 2013 Apr 3. PMID 23553151
- [Derived] Curtis PJ, Sampson M, Potter J, Dhatariya K, Kroon PA, Cassidy A. Chronic ingestion of flavan-3-ols and isoflavones improves insulin sensitivity and lipoprotein status and attenuates estimated 10-year CVD risk in medicated postmenopausal women with type 2 diabetes: a 1-year, double-blind, randomized, controlled trial. Diabetes Care. 2012 Feb;35(2):226-32. doi: 10.2337/dc11-1443. Epub 2012 Jan 16. PMID 22250063